CLINICAL TRIAL: NCT06659302
Title: Evaluating the Feasibility of a Virtual Stepped Mental Health Care Intervention for Children with Congenital Heart Disease
Brief Title: Feasibility of a Virtual Mental Health Intervention for Children with Congenital Heart Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: The Hospital for Sick Children (Other); Alberta Children's Hospital (Other)
Responsible Party: Principal Investigator, Marsha Vasserman, Pediatric Neuropsychologist, University of Calgary
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB24-1232
Record Dates: First submitted 2024-10-21; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Congenital Heart Disease (CHD)
Keywords: heart; CHD; behavior; family stress
MeSH Terms: conditions — Heart Defects, Congenital; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intro meeting (Experimental): Participants will be sent baseline questionnaires online through REDCap (Research Electronic Data Capture; see Appendix 1-email templates), a secure web application, and housed on a secure server. Participants will access a unique REDCap survey link via email to complete questionnaire measures after consenting to the study. After completion of the baseline questionnaires, participants will be connected with an I-InTERACT-North therapist for an Introductory Meeting to conduct a baseline elevation session. If participants do not wish to enroll in the full program, post-intervention questionnaires will be administered online through REDCap post step 1. If they wish to proceed to the full program, they will complete the questionnaires after step 2 or 3.
  Interventions: Behavioral: I-inTERACT North Step 1
- Two sessions (Experimental): Step 2: Parents who were identified as high stress/behaviour on the baseline questionnaires and/or based on the introduction meeting in Step 1, will be invited to participate in the initial two therapist-guided I-InTERACT-North sessions that focus on family stress and positive parenting strategies. Each session includes both an online psychoeducational module and a video conferencing session with a therapist. Session frequency is subject to change based on parent schedule preference and availability. Each session will last 60 minutes and will be video recorded (with consent from the participants). Sessions will be delivered to parents using Zoom, a secure online video conferencing platform (https://zoom.us/). If they wish to proceed to the full program, they will complete the questionnaires after step 3.
  Interventions: Behavioral: I-inTERACT North step 2
- Full Program (Experimental): Step 3: Families will be invited to participate in the full I-InTERACT-North program. The full program will provide an additional 5 online modules with live therapist videoconference coaching sessions. All sessions are strongly encouraged but for parents who do not complete the additional sessions, we will track what is completed and parents may still complete outcome measures. Based on previous work, average time of completion for the full program is 8-12 weeks. Each session will last 60 minutes and will be video recorded (with consent from the participants). Sessions will be delivered to parents using Zoom, a secure online video conferencing platform (https://zoom.us/). Before each session, parents will receive a meeting invitation link via email. After completing the program, participants will complete online questionnaires through REDCap. All participants will be invited to complete study follow-up questionnaires.
  Interventions: Behavioral: I-inTERACT North

INTERVENTIONS:
Behavioral: I-inTERACT North Step 1 — Initial questionnaires completed followed by initial meeting with therapist for baseline evaluation.
  Arms: Intro meeting
Behavioral: I-inTERACT North step 2 — Two online modules completed by family plus two online zoom coaching sessions with therapist.
  Arms: Two sessions
Behavioral: I-inTERACT North — Full program will consist of an additional 5 sessions with online modules and virtual coaching sessions with therapist.
  Arms: Full Program

SUMMARY:
Children with congenital heart disease are at much higher risk for behavioral and emotional difficulties in early childhood and beyond 1. However, intervention programs aimed at this population are limited and few have explored the efficacy of behavioral parent training on child behavior and parent stress in children with CHD. Few evidence-based behavior intervention programs are available in the community for families of children with CHD and behavioral struggles and many families struggle to stick with long-term treatment given the multiple appointments and responsibilities that are often already associated in parenting children with chronic health conditions. As such, more targeted, shorter and more accessible interventions are very needed. Established internet-based treatments such as I-InTERACT-North, are particularly well-suited for adaptation to stepped-care delivery due to prior implementation success, readily adaptable intensity of online content and therapist contact.

This study will evaluate whether I-InTERACT North is a feasible intervention to implement in a step-care model and whether it is acceptable to families and impacts behavior and family functioning.

DETAILED DESCRIPTION:
I-InTERACT-North was designed to be delivered online with a longstanding record of success in virtual service among children and families with behavioural challenges and parenting stress associated with acquired brain injury. The program contains key components that can be used in a stepped-care model to address parent stress and child behavioural concerns: 1) psychoeducation regarding the impact of heart disease on brain development, as well as behavior and emotion regulation skills in children, and 2) parenting strategies that foster responsiveness and consistency in the home. These two components have been shown to be effective in optimizing child behavior outcomes and reducing parental distress.

The program combines online learning modules with 1:1 parent-coaching provided in the family's home by videoconferencing. Coaching sessions reinforce content and provide direct live coaching on parent-responsivity skills. There is flexibility in when online modules are completed and video conference sessions are scheduled, essential considerations for families balancing simultaneous work and child-care demands. One of the co-investigators (Williams) recently completed an open-label pre-post pilot feasibility trial of the transdiagnostic program at SickKids among families following neonatal medical illness/injury, an important cause of early behaviour and emotional regulation issues, with promising implementation outcomes and preliminary indices of improvement in child behaviour and parent stress.15 In this study, approximately 69% of eligible families contacted consented; and 86% enrolled completed the 7-session program. Parents and therapists reported high overall satisfaction with the program (100%), including acceptability of both the online modules (95%) and the videoconference sessions (95%). Child behaviour (d=0.50, See Figure 1) and parenting confidence and skill (d = 0.45, 0.64) also improved. Among participants who did not complete the program, families cited lack of time as the number one barrier to participation. This stepped care approach directly addresses this concern by matching mental health services to the needs of families.

The current study leverages an existing evidenced-based virtual program (I-InTERACT-North) that contains key components to address stress and child behaviour concerns within a stepped-care model: 1) general psychoeducation regarding the impact of medical diagnosis on children and families, and 2) graduated intensity in coaching of parenting strategies that foster responsiveness, warmth and consistency in the home. These two components have longstanding effectiveness in optimizing child behavior and reducing parental distress.

Study Purpose and Objectives 2.1 Primary Objectives

1. To evaluate whether a stepped-care adaptation of I-InTERACT-North can be implemented as planned, measuring fidelity, acceptability, and engagement.
2. To assess accrual and dropout rates at each step.
3. To investigate program fidelity between our site and the main intervention site
4. To examine participant and care provider perceptions regarding intervention acceptability and satisfaction.
5. To evaluate the relationship between parent and child needs, key social demographic factors and program participation

Secondary Objectives

1) To measure the association between pre-and post-intervention short-term child behaviour and parent stress outcomes, parent responsivity and behavioural management skills, with hypothesized greater improvement following higher steps of engagement.

ELIGIBILITY:
Inclusion Criteria:

* Consent provided
* parent of a child aged 3 to 9 years,
* parent reported concerns regarding their child's externalizing behaviour
* child is followed in cardiology clinic at Alberta Children's Hospital.
* parent is able to speak and read English.

Exclusion Criteria:

* Child is outside of age range of the program (<3 or > 9 years of age)
* Significant major medical issues requiring ongoing inpatient care
* Currently participating in an equivalent family/parent therapy program (e.g., Incredible Years Parenting Program (IYPP), Positive Parenting Program (Triple P))
* Inability to read/write and communicate in English
* Inability to consent or complete study measures electronically (online)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Accrual Rate | 56 weeks from first participant contact
  the proportion of invited participants who consent to participate
Dropout Rate | 70 weeks after contacting first participant
  the proportion of participants who drop out of the study during Step 1, 2 or 3
Fidelity: | 70 weeks after contacting first participant
  the proportion of content covered from therapy protocols and questionnaires completed;
Acceptability & Satisfaction | 70 weeks after first participant contact
  the proportion of participants and therapists who rate the program as satisfactory or very satisfactory based on post-intervention; dropouts considered not-satisfied
Engagement & Adherence: | 70 weeks after first participant contact
  the amount of time (in hours/weeks) to complete intervention steps will be estimated by parents and therapists (for steps 2 and 3), the number of sessions completed an adherence index (sessions completed/total sessions scheduled)

SECONDARY OUTCOMES:
Child behavior concerns and intensity baseline | 1 day after signing consent
  Child behavior concerns and intensity will be measured using the Eyberg Child Behavior Inventory (ECBI), a 36-item checklist of mental health concerns. Following Step 1, reported elevated scores (T score>60) will be considered at-risk.
Parental stress baseline | 1 day after signing consent
  The Depression Anxiety and Stress Scale Short Form (DASS-21) will measure general distress in parents, with three subscales (depression, anxiety, and stress) with strong internal consistency, adequate construct validity and sensitivity to parent therapy; using cut-off scores of 60 for step 2
Child behavior at end of study | up to 25 weeks after signing consent
  ECBI will be used to measure child behavior concerns
Parent stress end of study | up to 25 weeks after signing consent
  DASS-21 will be used to measure parent stress

IPD SHARING:
Plan to Share IPD: Yes
deidentified fidelity data related to program implementation will be shared with Hospital for Sick Kids in Toronto who will be providing program support and supervision.

REFERENCES:
- [Background] Burek B, Ford MK, Hooper M, Green R, Kohut SA, Andrade BF, Ravi M, Sananes R, Desrocher M, Miller SP, Wade SL, Williams TS. Transdiagnostic feasibility trial of internet-based parenting intervention to reduce child behavioural difficulties associated with congenital and neonatal neurodevelopmental risk: introducing I-InTERACT-North. Clin Neuropsychol. 2021 Jul;35(5):1030-1052. doi: 10.1080/13854046.2020.1829071. Epub 2020 Oct 8. PMID 33028141
- [Background] Wiggins TL, Sofronoff K, Sanders MR. Pathways Triple P-positive parenting program: effects on parent-child relationships and child behavior problems. Fam Process. 2009 Dec;48(4):517-30. doi: 10.1111/j.1545-5300.2009.01299.x. PMID 19930436
- [Background] Masten AS, Hubbard JJ, Gest SD, Tellegen A, Garmezy N, Ramirez M. Competence in the context of adversity: pathways to resilience and maladaptation from childhood to late adolescence. Dev Psychopathol. 1999 Winter;11(1):143-69. doi: 10.1017/s0954579499001996. PMID 10208360
- [Background] Antonini TN, Raj SP, Oberjohn KS, Cassedy A, Makoroff KL, Fouladi M, Wade SL. A pilot randomized trial of an online parenting skills program for pediatric traumatic brain injury: improvements in parenting and child behavior. Behav Ther. 2014 Jul;45(4):455-68. doi: 10.1016/j.beth.2014.02.003. Epub 2014 Feb 13. PMID 24912459
- [Background] Cohen GH, Tamrakar S, Lowe S, Sampson L, Ettman C, Linas B, Ruggiero K, Galea S. Comparison of Simulated Treatment and Cost-effectiveness of a Stepped Care Case-Finding Intervention vs Usual Care for Posttraumatic Stress Disorder After a Natural Disaster. JAMA Psychiatry. 2017 Dec 1;74(12):1251-1258. doi: 10.1001/jamapsychiatry.2017.3037. PMID 28979968